CLINICAL TRIAL: NCT05135325
Title: Encouraging Blood Donation in Patients With a Blood Type in Short Supply
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2021-0476
Record Dates: First submitted 2021-11-15; First posted 2021-11-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Health Behavior
Keywords: Blood donations; Nudge; Behavior change
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The patients in the study will not know that other messages are being sent to other patients, although they will see the text of their own message. Providers will be blind to patient conditions.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- No-blood-type message (Experimental): This group will receive a message that does not mention the patient's blood type, or that the patient's blood type is in short supply.
  Interventions: Behavioral: Patient portal message
- Blood-type message (Experimental): This group will receive a message that mentions the patient's blood type and that states their blood type is in short supply.
  Interventions: Behavioral: Patient portal message; Behavioral: Social responsibility
- Shortage control (No Intervention): This group will not receive a message.
- No-shortage control (No Intervention): This group will not receive a message.

INTERVENTIONS:
Behavioral: Patient portal message — Portal message encourages patients to donate blood
  Arms: Blood-type message; No-blood-type message
Behavioral: Social responsibility — Message specifies that there is a shortage of the patient's blood type
  Arms: Blood-type message

SUMMARY:
As of November 2021, partly due to the COVID-19 pandemic, there has been a months-long national shortage of several types of blood in the U.S. (O-Pos, O-Neg, A-Neg, B-Neg, and AB-Neg), which has extended to a local blood shortage within the Geisinger community. The broad aim of this collaborative healthcare operations quality improvement project is to determine whether a message indicating that a patient's own blood type is in short supply increases the likelihood that they will donate, compared to a message that mentions a blood shortage without referencing the patient's blood type, or no message at all. Scientists in Geisinger's Behavioral Insights Team (BIT), part of Geisinger's Steele Institute for Health Innovation, will collaborate with Miller Keystone, where Geisinger refers patients who wish to donate blood and from whom Geisinger receives blood for clinical purposes. Patients with one of the needed blood types will be randomized to receive 1) a message about a blood shortage that does not specify the blood types in short supply or their own blood type (no-blood-type message), 2) the same message modified slightly to specify the recipient's blood type, and to mention that their blood type is in short supply (blood-type message), or 3) no message (shortage control group). A second no-contact control group of patients without any of the needed blood types will also be observed (no-shortage control group). Both the blood-type and no-blood-type messages are informed by behavioral science, emphasizing supply needs in local hospitals and providing community-relevant examples of why someone might need blood (e.g., farming or industrial accidents). The BIT will compare how many patients in each group choose to donate blood. They hypothesize that: 1) patients who receive either message will be more likely to donate than patients who receive no message; and 2) patients who receive the blood-type message will be more likely to donate than those who receive the no-blood-type message. With respect to the latter hypothesis, informing the recipient that they have one of the needed blood types may increase their perception that they are in a semi-unique position to help someone in need as compared to a more general message that may suffer from a diffusion of responsibility effect.

ELIGIBILITY:
Inclusion Criteria:

* Documented blood type in short supply (for message groups and shortage control group)
* Documented blood type not in short supply (for no-shortage control group)
* Age 18+

Exclusion Criteria:

* Hemoglobin test result < 12.5 within the 3 months prior to list creation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59093 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-06-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants Who Attended a Donation Appointment | Within 6 weeks of the final message send date
  Attended a donation appointment within 6 weeks of their message send date, regardless of whether they donated. This outcome includes patients who were unable to donate for any reason (e.g. low hemoglobin) or patients who showed up to the appointment but decided to leave before donating.

SECONDARY OUTCOMES:
Number of Participants Who Successfully Donated Blood | Within 6 weeks of the final message send date
  Attended a donation appointment within 6 weeks of their message send date and successfully donated, excluding patients who were turned away from or left their appointment without donating.
Number of Participants Who Scheduled a Blood Donation Appointment | Within 2 weeks of the final message send date
  Scheduled an appointment within 2 weeks of their message send date.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Goren, PhD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data with no personally identifiable information will be made available to other researchers on the Open Science Framework for transparency.
Supporting Information: Analytic Code
Time Frame: The data will become available after publication of study results in a scientific journal and will be available as long as the Open Science Framework hosts the data.
Access Criteria: The data on the Open Science Framework will be open to anyone requesting that information.
URL: http://osf.io

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/25/NCT05135325/SAP_001.pdf